CLINICAL TRIAL: NCT07276425
Title: Early and Long-term Clinical Efficacy and Local Tissue and Peripheral Immune Changes Following Dupilumab Treatment in Prurigo Nodularis Patients
Brief Title: Early and Long-Term Efficacy and Immune Changes With Dupilumab in Prurigo Nodularis
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Dr M.S. de Bruin-Weller, Professor, UMC Utrecht
Other Study IDs: 12-407; 2023ESR0000155 (Other: Sanofi)
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Prurigo Nodularis (PN)
Keywords: prurigo nodularis; dupilumab
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Biospecimen Retention: Samples With DNA — Blood samples and skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dupilumab — In the Netherlands, the standard care for patients with moderate-to-severe prurigo nodularis who have failed or are contraindicated to conventional systemic immunosuppressive treatments consists of 300 mg of dupilumab administered subcutaneously every two weeks, following a loading dose of 600 mg administered subcutaneously.
  Other Names: Dupixent

SUMMARY:
With the arrival of dupilumab as the first available targeted therapy for PN, there is an unmet need for real-world data and translational research on the working mechanism of dupilumab on PN, to optimize individualized targeted treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with moderate-to-severe prurigo nodularis starting dupilumab treatment

Exclusion Criteria:

* Unwilling to participate in the BioDay registry
* (For translational endpoints only) Unwilling to participate in UMC Utrecht Biobank

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary and tertiary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Peak Pruritus NRS (PP-NRS) | From enrollment to 52 weeks of treatment
  Peak pruritus NRS of the past 24 hours
Investigator Global Assessment scale of Prurigo Nodularis stage (IGA-PN) | From enrollment to 52 weeks of treatment
  Investigator Global Assessment scale of Prurigo Nodularis stage
Drug survival | From enrollment to 52 weeks of treatment
  Duration of dupilumab treatment, reasons for discontinuation
Adverse events | From enrollment to 52 weeks of treatment
  Data on the incidence, severity, relation to dupilumab and clinical consequences of adverse events
Skin homing T cell subtypes | Up to 52 weeks of treatment
Serum levels of relevant proteins | Up to 52 weeks of treatment
Systemic epigenetic changes | Up to 52 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No